CLINICAL TRIAL: NCT05080946
Title: Pilot Study to Assess the Efficacy of Aspirin to Improve Immunological Features of Ovarian Tumors
Brief Title: Using Aspirin to Improve Immunological Features of Ovarian Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Sharp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: MCC-20870; E01775.1a (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Participants Randomized to Aspirin (Experimental): Participants randomized to this arm will receive 325mg daily dose aspirin
  Interventions: Drug: Aspirin 325mg
- Participants Randomized to Placebo (Placebo Comparator): Participants randomized to this arm will receive a daily dose of a placebo (inactive substance)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin 325mg — Participants will receive a tablet of 325mg aspirin that is taken once daily by mouth. Study treatment begins on first day of neoadjuvant chemotherapy for up to 5 "cycles". Participants will be expected to take the study treatment for between 63 and 175 days (3-5 cycles). Participants will stop taking study treatment 7 days prior to participants interval debulking surgery.
  Arms: Participants Randomized to Aspirin
Drug: Placebo — Participants will receive a placebo tablet that is taken once daily by mouth. Study treatment begins on first day of neoadjuvant chemotherapy for up to 5 "cycles". Participants will be expected to take the study treatment for between 63 and 175 days (3-5 cycles). Participants will stop taking study treatment 7 days prior to participants interval debulking surgery.
  Arms: Participants Randomized to Placebo

SUMMARY:
The purpose of the study is to evaluate the effectiveness of aspirin with neoadjuvant chemotherapy for decreasing markers of immune suppression in the tumor at interval debulking surgery, in women with diagnosed ovarian, fallopian tube, or peritoneal carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Participants that are greater than or equal to 18 years of age
* For U.S. sites, patients can read and understand English or Spanish; for Canadian site, participants can read and understand English or French
* Histology confirmed, or clinical suspicion of, invasive epithelial ovarian, fallopian tube, or peritoneal carcinoma. Must be grade 2 or 3 or high (where high is defined as grade 2/3). All histologies including serous, endometrioid, clear cell sarcoma, or carcinosarcoma histology is acceptable. Mixed histology also acceptable.
* Treatment naïve for this cancer diagnosis
* Planned for neoadjuvant chemotherapy (platinum-based doublet with taxane +/- anti-VEGF antibody) for at least 3 but no more than 5 cycles followed by an interval debulking surgery. [Note: this study evaluates response while on neoadjuvant treatment. The final collection of specimen and questionnaire is at the time of surgery and immediate post-operative state. Therefore, there are no eligibility criteria related to treatment in the adjuvant setting (e.g., intraperitoneal treatment) and adjuvant therapy should proceed as the physician deems appropriate.]
* Measurable disease as defined by RECIST 1.1, CT scan (with or without contrast) within 12 weeks of study enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1, or 2
* Able to provide tissue biopsy (core or excisional) sufficient for diagnosis and biomarker analysis, may use outside archival tissue if available.
* If currently using anti-coagulation medication, no contraindication for temporary stoppage of use during the study based on physician judgement
* Willing and able to swallow pills without difficulty
* Un-transfused platelet count > 100,000 cells/μL
* Willing and able to participate in all required evaluations and procedures in this study protocol (e.g. undergoing treatment, scheduled visits and examinations, serum testing, questionnaires, pill log/diary)
* Absolute neutrophil count > 1.5 x 109 cells/L
* Hemoglobin > 9.0 g/dL, may use transfusions and the value can be post-transfusion
* Estimated creatinine clearance of > 30 mL/min, calculated using the formula Cockcroft-Gault [(140-age) x Mass (kg)/(72 x creatinine mg/dL)] x 0.85 for female
* No severe hepatic impairment defined as AST or ALT elevation < 2.5 x institutional ULN, unless liver metastasis is present < 5 x ULN

Exclusion Criteria:

* Definite contraindication for either aspirin use or stopping current aspirin use based on physician's clinical judgment
* History of vascular event in the last 12 months (e.g., myocardial infarction or unstable angina, stroke, coronary artery angioplasty or stenting, coronary artery bypass graft, relevant [serious or significant] arrhythmias, significant vascular disease, congestive heart failure or vascular interventions).
* History of hypertensive crisis and/ or uncontrolled HTN, systolic blood pressure > 150 mmHg; diastolic blood pressure > 90mmHg. Participants must have blood pressure < 150/90 mmHg taken in a clinic setting by a medical professional within 2 weeks prior to starting study.
* Current or history of ulcers which prohibits aspirin consumption, severe hepatic failure, or acute or chronic renal disease where aspirin use is contraindicated
* History of gastrointestinal or genitourinary bleeding or other bleeding diathesis or coagulopathy within 6 months prior to enrollment of study
* Uncontrolled erosive esophagitis requiring 2 or more treatments
* Other cancer diagnosis in the last 3 years other than non-melanoma skin cancer
* Autoimmune disorder requiring systemic therapy
* Chronic steroid use defined as 3 weeks in the past year or any length of time in the past 30 days.
* Other aspirin or NSAID hypersensitivities or contraindications (e.g. allergy)
* History of bariatric surgery
* Currently pregnant at the Screening visit or planning on becoming pregnant during the study period
* Participant is unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with study medication.
* Metabolism CYP2C9, known G6PD deficient patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in intratumoral density of immunosuppressive T-regulatory (FOXP3+) cells from diagnostic biopsy to interval debulking surgery | Up to 5 months
  Change in intratumoral density of immunosuppressive T-regulatory (FOXP3+) cells will be measured by using this formula: (density in the debulking surgery tissue sample - density in the biopsy tissue sample)*100 / density in the biopsy tissue sample.
Change in intratumoral density of M2 tumor-associated macrophages (CD163+ cells) from diagnostic biopsy to interval debulking surgery | Up to 5 Months
  Change in intratumoral density of of M2 tumor-associated macrophages (CD163+ cells) will be measured by using this formula: (density in the debulking surgery tissue sample - density in the biopsy tissue sample)*100 / density in the biopsy tissue sample.

SECONDARY OUTCOMES:
Change in density of tumor COX1 | Up to 5 Months
  Change in density of tumor COX1 will be measured by using this formula: (density in the debulking surgery tissue sample - density in the biopsy tissue sample)*100 / density in the biopsy tissue sample.
Change in density of tumor COX2 | Up to 5 Months
  Change in density of tumor COX2 will be measured by using this formula: (density in the debulking surgery tissue sample - density in the biopsy tissue sample)*100 / density in the biopsy tissue sample.
Change in blood levels of IL-6 | Up to 84 days
  Investigators will calculate the percent change in the concentration of the biomarker from baseline to Visit 4
Change in blood levels of p-selectin | Up to 84 days
  Investigators will calculate the percent change in the concentration of the biomarker from baseline to Visit 4
Change in blood levels of CA 125 | Up to 84 days
  Investigators will calculate the percent change in the concentration of the biomarker from baseline to Visit 4
Change in tumor burden as defined by RECIST 1.1 | Up to 5 Months
  Change in tumor burden be assessed using Response Evaluation Criteria in Solid Tumors guideline version 1.1 (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Yi Chern, MD, Principal Investigator — Moffitt Cancer Center
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - Oregon Health and Science University, Portland, Oregon
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Clinical Trial Search — https://moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE